CLINICAL TRIAL: NCT04698954
Title: Evaluation of the Adapted Adherence Improving Self-Management Strategy Intervention in Chronic Heart Failure Patients - a Randomized Controlled Trial
Brief Title: Evaluating the Adherence Improving Self-Management Strategy Intervention in Chronic Heart Failure Patients
Acronym: AIMS-CHF RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Maas Hospital Pantein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL74248.091.20
Record Dates: First submitted 2020-12-14; First posted 2021-01-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2020-12

CONDITIONS: Chronic Heart Failure; Heart Decompensation; Myocardial Failure; Preserved Ejection Fraction; Reduced Ejection Fraction
Keywords: Medication adherence; Physical activity; Step count; Self-management; Behavioural intervention; Self-care; Symptom monitoring; Symptom management; Electronic monitoring
MeSH Terms: conditions — Heart Failure; Medication Adherence; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIMS intervention group (Experimental): A nurse-delivered behavioural intervention focussing on medication adherence, physical activity, and symptom management integrated in routine clinical care. AIMS-CHF incorporates nurse-counselling and feedback from electronic monitoring of medication use (using MEMS-buttons) and physical activity (using pedometers).
  Interventions: Behavioral: Adherence Improving self-Management Strategy
- Treatment-as-usual group (Active Comparator): Participants in the control group will receive treatment as usual. They will visit the out patient clinic each 3 or 6 months for 30 minutes.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Behavioral: Adherence Improving self-Management Strategy — The AIMS intervention is a conversation between a patient and a trained nurse, imbedded in the usual care. It consists of structured modules with visual materials, developed based on a sound understanding of the factors that drive non-adherence and potent behaviour change techniques to modify those. These modules aim to enhance patient knowledge, motivation, self-efficacy, and skills for self-managing their treatment. As part of the intervention, patients use electronic monitors to track their own behaviour, namely a medication and a physical activity monitor. Together with the nurse they examine these results to identify adherence problems and solutions and make a plan.
  Arms: AIMS intervention group
Other: Treatment-as-usual — Participants in the control group will receive treatment as usual. They will visit the nurse in the out patient clinic each 3 or 6 months for 30 minutes.
  Arms: Treatment-as-usual group

SUMMARY:
Patient non-adherence to treatment recommendations is common and decreases the effectiveness of Chronic Heart Failure (CHF) treatment. Improving adherence towards medication intake, physical activity, symptom monitoring/management might prolong life, alleviates symptoms, increases quality of life, and reduces hospital admissions. The Adherence Improving self-management Strategy (AIMS) is a nurse delivered intervention, integrated in routine clinical care, aiming to better support patients in their treatment. AIMS has previously been demonstrated to be (cost) effective amongst HIV patients. Based on the literature and advisory boards with healthcare providers and CHF patients, AIMS is adapted to CHF (AIMS-CHF).

The aim of the study is to evaluate the effectiveness of the AIMS intervention on adherence regarding medication, physical activity, and symptom management compared to treatment-as-usual in patients with chronic heart failure.

DETAILED DESCRIPTION:
◦Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.

Data for the primary outcome medication adherence will be monitored electronically and data will be downloaded during regular clinic visits and automatically downloaded to a protected study server. The quality of electronically monitored medication adherence data depends on whether the electronic monitors are used adequately. The research team will monitor adequate use of these electronic monitors at the start of the study.

Data for secondary outcomes will be collected through questionnaires and the research team will follow-up on participants not completing those. Statistical analysis plans will be uploaded before data collection is completed and the database is accessed.

◦Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

The quality of electronically monitored medication adherence data depends on whether the electronic monitors are used adequately. At study exit, data will be discussed with all patients. When electronic monitoring data is completely missing or suggests very low adherence (depending on the sample distributions, but this could be e.g., <50% of doses taken) in the presence of well-controlled symptoms; and the participant self-reports poor use of the electronic monitor, then a sensitivity analysis will be conducted with those electronic monitoring data replaced by the participants' self-reported adherence.

Physical activity, will be self-reported. The validity of this self-report will be examined against electronic physical activity measures used by participants in the treatment arm.

◦Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (for example, medical records, paper or electronic case report forms, or interactive voice response systems).

Not applicable

◦Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used (for example, World Health Organization Drug Dictionary, MedDRA), and normal ranges if relevant.

Not applicable

◦Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

Patient recruitment Heart failure patients in outpatient clinic will be approached by the health care professional to inform them about the study and subsequently an information letter will be handed over. This letter contains information concerning the nature, purpose and duration of the study as well as possible objections, risks of participation and the possibility to withdrawal at any time without the need to specify the reason. Subsequently, the treating physician, or the researcher, will explain all study procedures and answer any questions. In case the patient is willing to participate and deemed eligible, he/she is asked to sign the informed consent form, preferably in presence of their partner, family member or friend.

Data will be handled confidentially and will not be distributed to third parties. After informed consent, each participant will be given a unique code consisting of letters (the code name of the study) and a number (e.g. 001). The key linking to the patient identity will be stored in a secured file and only the involved investigators will have access to this key. Personal data will be handled in accordance with the Dutch Personal Data Protection Act. The research data will be stored for 15 years after finalisation of the project. The data required for the trail will be collected and stored in the electronic Case Report Form (eCRF) using Castor (Castor EDC 2019.1.15 or further, Ciwit B.V., The Netherlands) and afterwards exported to SPSS statistics 25 or R for the analyses. Only the involved investigators will have unrestricted access to all pseudonymized data. Patients in the intervention group will monitor their behaviour. For medication adherence applies each time they open the MEMS bottle or push the button the date will be registered. The MEMS cap is ISO 9001 certified, CE-marked, HIPPA compatible, compliant with FDA 21 CFR part 11 and GDPR compliant. Stored information can be transferred at any time through the MEMS Reader to the MEMS adherence software for immediate analysis and interpretation. The data transmission can be done using a dedicated MEMS USB NFC reader. The data is securely transferred and stored encrypted on AARDEX servers using end-to-end encryption. Data storage is secured by continuous backups and data replication. The data is only accessible when logging in with the correct credentials (login/email and password), and only be accessible for the HCP (direct feedback) and the researcher (data analysis).

For the activity tracker applies the following; the data from the activity tracker is in the possession of the patient itself, and will share these data with the HCP. During wear-time, the activity tracker continuously collects data about the stepping, time of the patient. Data collection and storage of the activity tracker is GDPR compliant and data is stored on secure servers protected with pseudonymization and encryption.

Study related correspondence, signed Informed Consent forms, and source documents are to be maintained by the study site and archived in a locked cabinet for a minimum of 15 years after the end of this study. Source data will be entered at worksheets in the eCRF and afterwards exported to SPSS statistics 25 or R for the analyses.

* Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.

  136 patients will be recruited (based on a Sample size calculation: effect size: 0.5223; 1-β=0.80; α=0.05, and assuming a 15% dropout).
* Plan for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Depending on the type of missingness (e.g., at random, completely at random) appropriate data imputation procedures will be used if no alternative data sources for the missing datapoint is available

◦Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

Primary outcome variable Linear mixed-effects models will be used to assess the effects of AIMS-HF versus treatment-as-usual on dosing adherence measured with MEMS. Baseline dosing adherence will be used as covariate and intervention assignment as the treatment variable (0/1). Mean dosing compliance will be calculated per 3-month period and included as repeated time points.

Secondary study parameter(s) Regression analyses will be conducted for the secondary outcomes (questionnaires), where the baseline value of the dependent variables and the treatment variable (0/1) are included as the predictors.

Tertiary study parameter(s) To explore the effects on event-free survival (time to the first event) Kaplan-Meier survival analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Chronic Heart Failure (from either preserved or non-preserved systolic functions)
* New York Heart Association class II and III
* Able to understand and perform study related procedures
* Has an appointment at the HF clinic of at least once per 6 months

Exclusion Criteria:

* Unable to give informed consent
* New York Heart Association class I or IV
* Participation in another interventional study targeting medication adherence, physical activity, symptom monitoring, and/or diet.
* A coexisting imminently terminal illness, such as cancer or chronic renal failure requiring dialysis.
* Patients in titration phase (due to multiple changes in medication regimen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  Medication will be objectively assessed by a medication registration button, which is a medication event monitoring system (MEMS). The percentage of days with the correct amount of intakes, indicates the dosing adherence.

SECONDARY OUTCOMES:
Physical activity (SQUASH) | Change from baseline, at 6 and 12 months follow-up
  Physical activity will be measured subjectively, using the Short Questionnaire to Assess Health (SQUASH) consisting of 11 items.
Physical activity (SBQ) | Change from baseline, at 6 and 12 months follow-up
  Physical activity will be measured subjectively, using Sedentary Behaviour Questionnaire (SBQ), consisting of 9 items.
Physical activity (Garmin Vivofit 4) - number of steps | Change from baseline (2 weeks prior intervention consult at 6 months), at 9 and 12 months follow up
  Physical activity will also be measured objectively (intervention group only), by the Garmin Vivofit 4. It registers the number of steps taken each day.
Physical activity (Garmin Vivofit 4) - active minutes | Change from baseline (2 weeks prior intervention consult at 6 months), at 9 and 12 months follow up
  Physical activity will also be measured objectively (intervention group only), by the Garmin Vivofit 4. It registers active minutes each day.
Physical activity (Garmin Vivofit 4)- moving distance | Change from baseline (2 weeks prior intervention consult at 6 months), at 9 and 12 months follow up
  Physical activity will also be measured objectively (intervention group only), by the Garmin Vivofit 4. It registers moving distance each day.
Heart failure self-care | Change from baseline, at 6 and 12 months follow-up
  The valid Self-Care of Heart Failure Index (SCHFI) is a 15-item questionnaire developed to get insight in the patients' ability to perform the specific HF self-care behaviours, including symptom monitoring/management.
Self-management | Change from baseline at 12 months follow-up
  The American short form Patient Activation Measure (PAM) is a 13-item instrument which assesses patient (or consumer) self-reported knowledge, skills, and confidence for self-management of one's health or chronic condition.
Health related quality of life | Change from baseline at 12 months follow-up
  The health related quality of life questionnaire for patients with heart failure is the 21-item Minnesota Living with Heart Failure Questionnaire (MLHFQ).

OTHER OUTCOMES:
Cardiac Event Free Survival | Up to 1 year and 5 years follow up
  This is a composite measure of cardiac events (cardiac related hospitalization, cardiac related emergency department visit or cardiac related death)

CONTACTS AND LOCATIONS:
Overall Officials: Marijn de Bruin, prof. dr., Principal Investigator — Radboudumc, RIHS, IQ Healthcare
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - CWZ, Nijmegen, Gelderland
  - Maasziekenhuis Pantein, Beugen, North Brabant

IPD SHARING:
Plan to Share IPD: Undecided